CLINICAL TRIAL: NCT04728178
Title: Comparison of Perioperative Standard Fluid Management and Goal-Directed Fluid Management in Patients Undergoing Head and Neck Surgery: A Prospective Randomized Clinical Trial
Brief Title: Comparison of Perioperative Standard Fluid Management and Goal-Directed Fluid Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Demet Altun, attending anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1122
Record Dates: First submitted 2021-01-20; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Perioperative Fluid Management
Keywords: fluid therapy; prolonged oxygen demand; perioperative fluid balance
MeSH Terms: interventions — Crystalloid Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): In the control group, fluid management was set as MAP (Mean arterial pressure) 65 mmHg and above and diuresis 0.5ml/kg/hour and above. Crystalloid infusion at 7ml/kg/hour was started. When SVV value increased to 13% and over in the study group, 250 ml of crystalloid was given in the first stage, and if it continued to be 13% and over, 250 ml of colloid bolus was given. Vasoconstrictor agent was used when SVV was below 13% and MAP was below 65 mmHg.
  Interventions: Other: Crystalloid solution; Other: Colloid solution
- control group (Placebo Comparator): In the control group, fluid management was set as MAP (Mean arterial pressure) 65 mmHg and above and diuresis 0.5ml/kg/hour and above. Crystalloid infusion at 7ml/kg/hour was started. They were given 250 ml of crystalloid in the first stage if the MAP was below 65 mmHg, and 250 ml of colloid bolus if the hypotensive episode continued. If hypotension persisted despite these fluid boluses, a vasoconstrictor agent was used. In addition, when the diuresis of the patients was detected at 0.5mg/kg/hr or less, 250 ml of colloid bolus was administered.
  Interventions: Other: Crystalloid solution; Other: Colloid solution

INTERVENTIONS:
Other: Crystalloid solution — Crystalloid solution is a true solution and is able to pass through a semipermeable membrane.
Other: Colloid solution — Colloid solution is a heterogeneous mixture whose particle size is intermediate between those of a solution and a suspension.

SUMMARY:
To compare the goal-directed fluid therapy based on the data obtained from the hemodynamic monitoring system, which provides continuous CO, SV and SVV measurements through arterial pressure wave with standard fluid therapy in perioperative fluid management of patients undergoing head and neck surgery.

DETAILED DESCRIPTION:
Following the ethics committee approval and patients consent, the study was completed with a total of ASA I-III, 60 patients over the age of 18 who will undergo head and neck surgery.After randomization, patients underwent arterial cannulation. The arterial cannulas of the study group patients were integrated into the hemodynamic monitoring system with a special transducer, and their fluid management was planned to achieve a target value of 13% or less through SVV monitoring. In the control group, fluid management was set as MAP (Mean arterial pressure) 65 mmHg and above and diuresis 0.5ml/kg/hour and above. Crystalloid infusion at 7ml/kg/hour was started in both groups. When SVV value increased to 13% and over in the study group, 250 ml of crystalloid was given in the first stage, and if it continued to be 13% and over, 250 ml of colloid bolus was given. Vasoconstrictor agent was used when SVV was below 13% and MAP was below 65 mmHg. The patients in the control group were given 250 ml of crystalloid in the first stage if the MAP was below 65 mmHg, and 250 ml of colloid bolus if the hypotensive episode continued. If hypotension persisted despite these fluid boluses, a vasoconstrictor agent was used. In addition, when the diuresis of the patients was detected at 0.5mg/kg/hr or less, 250 ml of colloid bolus was administered.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the study
2. ASA classification 1, 2 or 3
3. The patients who will undergo head and neck surgery

Exclusion Criteria:

1. Being under the age of 18 or over the age of 80
2. Presence of serious cardiac, renal and liver pathology ( ejection fraction< %35 and/or glomerular filtration rate< 30ml/kg/min, kreatinin>2,5mg/dl and/or abnormal liver function test)
3. The patients who have heart rhythm problems such as atrial fibrillation, sinus tachycardia, ventricular extrasystoles
4. The patients who have a peripheral arterial disease
5. Being a morbid obese ( BMI>40 kg/m2)
6. the patients who may have considered difficult airway

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative fluid balance | during surgery
  the total and additional amount of crystalloid and colloid fluid fluid given during the surgery

SECONDARY OUTCOMES:
Prolonged IMV demand | during 8 hours after surgery
  The need for artificial respiration for 8 hours or more in patients admitted to the postoperative intensive care unit.
Prolonged oxygen demand | during 8 hours after surgery
  The need for additional oxygen application with a mask for 8 hours or more in patients who are taken into postoperative service follow-up.
Heart rate | during surgery
  EKG
Blood Pressure | during surgery
  Arterial line and pressure transducer
hospitalisation time | postoperative period (up to 6 weeks)
  calendar
lenght of stay in ICU | postoperative period (up to 6 weeks)
  calendar
hypoxia | during surgery
  blood gas machine
hypercarbia | during surgery
  blood gas machine
pulmonary infection | postoperative period (up to 6 weeks)
  sputum culture test

CONTACTS AND LOCATIONS:
Overall Officials: Demet Altun Bingol, Assoc. Prof., Principal Investigator — Istanbul University; Nuray Turkut, MD, Principal Investigator — Istanbul University; Cansu Uzuntürk, Resident, Principal Investigator — Istanbul University; Emre Çamcı, Prof., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Davies SJ, Minhas S, Wilson RJ, Yates D, Howell SJ. Comparison of stroke volume and fluid responsiveness measurements in commonly used technologies for goal-directed therapy. J Clin Anesth. 2013 Sep;25(6):466-74. doi: 10.1016/j.jclinane.2013.04.010. Epub 2013 Aug 17. PMID 23965199
- [Background] Funk D, Bohn J, Mutch W, Hayakawa T, Buchel EW. Goal-directed fluid therapy for microvascular free flap reconstruction following mastectomy: A pilot study. Plast Surg (Oakv). 2015 Winter;23(4):231-4. doi: 10.4172/plastic-surgery.1000937. PMID 26665136